CLINICAL TRIAL: NCT04349189
Title: Venous Thrombosis Biomarkers in Sickle Cell Disease and Sickle Cell Trait
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200068; 20-H-0068
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07-22

CONDITIONS: Sickle Cell Disease; Venous Thrombosis; Sickle Cell Trait; Hypercoagulable State; Venous Thromboembolism
Keywords: hypercoagulable state; Recurrence; Biomarkers; Venous Thromboembolism; Vascular Mortality; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell; Venous Thrombosis; Sickle Cell Trait; Thrombophilia; Venous Thromboembolism; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: 50 Men and Women with sickle cell disease and VTE
- Group 2: 50 Men and Women with sickle cell disease but no VTE
- Group 3: 50 Men and Women with sickle cell trait
- Group 4: 50 ethnically matched Men and Women without sickle cell disease, sickle cell trait, or VTE

SUMMARY:
Background:

Venous thromboembolism (VTE) includes the abnormal clotting of blood in a deep vein of the upper or lower limbs (deep vein thrombosis) that may travel to and block a blood vessel in the lung (pulmonary embolism). Some people with sickle cell disease (SCD)-a red blood cell disorder-seem to be at greater risk for developing these blood clots. Researchers want to study the blood of people with SCD and VTE as well as healthy people to develop better treatments to prevent blood clots.

Objective:

To study blood clotting in SCD because it is the most common cause of vascular death after a heart attack or stroke.

Eligibility:

People ages 18-80 who have SCD (with or without a history of blood clots) or the trait for SCD, and healthy volunteers

Design:

Participants will be screened with medical history, physical exam, and medical records review. They will give blood samples.

Participants will have phone calls either every 3 months or once a year, for 2 years. They will give updates on their health. They may give additional medical records. The phone calls may last up to 30 minutes.

If participants have a VTE or pain crisis episode, they may visit the Clinical Center. These visits may last up to 4 hours. They will repeat the screening tests and give blood samples.

Some participants may be invited to take part in blood studies.

After 2 years, some participants will have a follow-up visit at the Clinical Center.

Participation will last for about 2 years.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) the third most frequent cause of vascular mortality after myocardial infarction and stroke, occurs more frequently among Americans of African descent compared with other ethnic minorities in the US. VTEs are provoked by diverse risk factors but can be unprovoked in individuals with a hypercoagulable state, in whom there is a predisposition for thrombosis. Patients with Sickle Cell Disease (SCD) have added risk of VTE as the disease itself is a hypercoagulable state. VTE frequency is increased across the entire spectrum of SCD severity, in those experiencing both mild (HbSC patients) and severe sickling symptoms (HbSS/HbSbeta0 thalassemia patients). Studies show that up to 12% of patients with SCD have VTE events [deep vein thrombus (DVT) or pulmonary embolism (PE) or both] early in life by age 40, most of which are unprovoked. Moreover, owing to a persistent hypercoagulable state, SCD patients are at an unacceptably high risk for recurrence, particularly those in whom VTE was unprovoked. SCD patients who develop a VTE have a 24.1% risk of recurrence over 5 years. A history of a VTE in SCD is associated with greater mortality risk (Odd Ratio, OR = 2.88; Confidence Interval, CI = 2.35 - 3.52).

Our overall hypothesis is that the proinflammatory state associated with SCD perturbs the coagulation system and contributes to the thrombotic vascular pathobiology of SCD. Abnormal intravascular tissue factor expressed on monocytes and endothelial cells and circulating tissue factor positive extracellular vesicles released by these cells drive coagulation activation in SCD. Specifically, intravascular tissue factor forms the tenase complex (TF:VIIa) which converts factor X to factor Xa, generating the initial thrombin burst that possibly triggers intravascular thrombosis. Besides, heightened tissue factor exposure during acute sickling crises, increased release of tissue factor positive extracellular vesicles and inadequate clearance of the latter favors thrombin generation, fibrin deposition and thrombosis in the venous vasculature. SCD patients with VTE and/or recurrent VTE are therefore more likely to have more tissue factor positive extracellular vesicles and plasma tissue factor procoagulant activity compared with SCD patients without VTE.

Prospective cohort studies of extended duration/indefinite anticoagulation in non-SCD patients with an underlying hypercoagulable state have effectively reduced recurrence rates. However, similar studies of extended duration anticoagulation in SCD patients are lacking. Besides, whether exposing SCD patients to extended/indefinite anticoagulation increases bleeding risk to unacceptably high levels is unknown. Studying thrombogenic risk and specifically identifying those SCD patients who are at greatest risk for VTE recurrence therefore becomes a high priority. In addition, individuals with sickle cell trait are prone to thrombosis but few studies evaluate markers of thrombotic risk in these individuals. Such studies could provide a rationale for targeted primary or secondary VTE prophylaxis.

In the current proposal we will test the hypothesis that plasma tissue factor positive extracellular vesicles and tissue factor activity are elevated among SCD patients with VTE compared with SCD patients without VTE and in individuals with Sickle Cell Trait compared with ethnically matched controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

Sickle cell disease with and without VTE

* Sickle cell disease (HbSS, HbSC and HbS/beta-thalassemia genotypes) in steady state.
* Diagnosis of at least one or more VTE within 5 years of study enrolment confirmed by radiologic imaging (for SCD patients with VTE).
* Absence of clinical history of VTE (for SCD controls)
* Between 18 and 80 years of age.
* Ability to provide informed written consent.

Sickle cell trait

* Sickle cell disease (HbAS genotype).
* Absence of clinical history of VTE
* Between 18 and 80 years of age.
* Ability to provide informed written consent.

Ethnically matched controls

* Between 18 and 80 years of age.
* African, or of African descent.
* Ability to provide informed written consent.
* Absence of clinical history of VTE

EXCLUSION CRITERIA:

SCD with and without VTE

* Pregnancy (test done at enrollment; if a subject becomes pregnant during the study period, samples will not be obtained while the subject is pregnant and the subject will be taken off study).
* Patients on exchange transfusion or having received a simple blood transfusion in the past 60 days.
* Active viral infection as evidenced by testing positive for hepatitis B surface antigen or hepatitis C virus (HCV) antibody (Ab) with signs of active hepatitis B or C virus infection. If the subject is positive for HCV Ab, a reverse transcriptasepolymerase chain reaction test will be conducted. Subjects with hepatitis C may be rescreened after receiving appropriate hepatitis C treatment.
* Testing positive for human immunodeficiency virus 1 or 2 Ab with evidence for ongoing active infection (i.e., CD 4 count <400/microL and viral load >100,000 copies/ml) on antiretroviral therapy.
* Active acute inflammatory disorders rheumatoid arthritis or systemic lupus erythematosus on disease modifying therapy.
* Diabetes mellitus judged to be under poor control by the Investigator evidenced by a single fasting sugar value >250gm/dl or requiring >3 antidiabetic agents, including insulin (all insulins are considered 1 agent); use of insulin per se is not exclusionary.

SCT and ethnically matched controls

* Diagnosis of any of the following chronic disease or conditions: Sickle cell disease (HbSS, HbSC and HbS/beta-thalassemia genotypes).
* Clinical history of VTE.
* Pregnancy (test done at enrollment; if a subject becomes pregnant during the study period, samples will not be obtained while the subject is pregnant and the subject will be taken off study.
* Active viral infection as evidenced by testing positive for hepatitis B surface antigen or hepatitis C virus (HCV) antibody (Ab) with signs of active hepatitis B or C virus infection. If the subject is positive for HCV Ab, a reverse transcriptasepolymerase chain reaction test will be conducted. Subjects with hepatitis C may be rescreened after receiving appropriate hepatitis C treatment.
* Testing positive for human immunodeficiency virus 1 or 2 Ab with evidence for ongoing active infection (i.e., CD 4 count <400/microL and viral load >100,000 copies/ml) on antiretroviral therapy.
* Active acute inflammatory disorders rheumatoid arthritis or systemic lupus erythematosus on disease modifying therapy.
* Diabetes mellitus judged to be under poor control by the Investigator evidenced by a single fasting sugar value >250gm/dl or requiring >3 antidiabetic agents, including insulin (all insulins are considered 1 agent); use of insulin per se is not exclusionary.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The natural history of SCD 04-H-0161 protocol (NCT00081523) will specifically be leveraged to recruit participants with VTE. In this study we will assess feasibility of establishing a prospective natural history study of thrombosis in SCD. Establishing feasibility could lead to recruitment of SCD patients experiencing thrombosis, particularly those that are understudied including patients with HbSC disease.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
tissue factor positive | At baseline during study
  Number of tissue factor positive EVs/ml of plasma

CONTACTS AND LOCATIONS:
Overall Officials: Arun S Shet, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-H-0068.html

DOCUMENTS (1):
  • Informed Consent Form (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT04349189/ICF_000.pdf